CLINICAL TRIAL: NCT05190081
Title: Investigation Of the Effects Of Dual-Task And Single-Task Training In Older Adults With Age-Related Hearing Loss
Brief Title: Task Training In Older Adults With Age-Related Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, HANDE USTA, Doctor, Research Assisstant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 60116787-020/1933.
Record Dates: First submitted 2021-11-06; First posted 2022-01-13 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Hearing Loss; Age Related Hearing Loss; Physical Disability; Vestibular Disease
Keywords: Age Related Hearing Loss; Dual Task; Cognitive Function; Physical Function
MeSH Terms: conditions — Hearing Loss; Presbycusis; Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Intervention groups were formed as single-task training, dual-task training, and control group. Distribution was made into groups using a simple randomized number selection technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single-task training group (Experimental): Tasks were completed separately in the single-task training group
  Interventions: Other: TASK TRAINING
- dual-task training group (Experimental): Tasks were completed at the same time in the dual-task training group
  Interventions: Other: TASK TRAINING
- control group (No Intervention): No intervention was performed in the control group

INTERVENTIONS:
Other: TASK TRAINING — A special program including motor and cognitive tasks was prepared. Both lower and upper extremity motor tasks and verbal, arithmetic, auditory, and visual cognitive tasks were planned based on evidence. The dual-task and single-task training were held 2 days a week, 40 minutes, for a total of 10 sessions for 5 weeks. A patient-appropriate task was selected for each cognitive task each week.
  Arms: dual-task training group; single-task training group

SUMMARY:
This study aimed to examine the effects of single and dual-task training on physical function, cognitive function, quality of life, balance, concerns about falling, and activities of daily living in the elderly with age-related hearing loss.

The elderly who were diagnosed with age-related hearing loss in Pamukkale University Health, Practice and Research Center, Department of Otorhinolaryngology participated in the study. The elderly were allocated a single-task training group, dual-task training group, and control group. Thirteen patients in the single-task training group, 15 patients in the dual-task training group, 14 patients in the control group completed the study. Degrees of hearing loss were determined by pure tone audiometry. Evaluations, Senior Fitness Test, Montreal Cognitive Assessment, World Health Organization- Quality of Life- Old Module, Berg Balance Scale, Falls Efficacy Scale International, Functional Independence Measure, Dual Task Questionnaire, Dual Task Effect, were performed initially, after the interventions and at the 6th month. The interventions were carried out two days a week and 40 minutes, for five weeks.

DETAILED DESCRIPTION:
Outcome Measures Physical function, cognitive function, auditory function, quality of life, balance, concerns about falling, independence in activities of daily living, and dual-task performance were evaluated. Older adults were evaluated initially, after the dual-task and single-task training, and at 6th month for long-term control. All evaluations and interventions were carried out in an isolated and quiet environment in the examination room of the Department of Otorhinolaryngology.

Interventions A special program including motor and cognitive tasks was prepared. Both lower and upper extremity motor tasks and verbal, arithmetic, auditory, and visual cognitive tasks were planned based on evidence. Tasks were completed at the same time in the dual-task training group, were completed separately in the single-task training group. No intervention was performed in the control group. The dual-task and single-task training were held 2 days a week, 40 minutes, for a total of 10 sessions for 5 weeks. A patient-appropriate task was selected for each cognitive task each week. It has been tried to prevent the learning effect by providing individual and weekly progress according to the patients' performance in the tasks in the motor and cognitive parts. Variable priority instructions were used in the dual-task training group, and fixed priority instructions were used in the single-task training group. At the beginning and end of the intervention programs, 7 types of warm-up and cool-down exercises involving large muscle groups were performed for 10-minutes. Each task in the intervention programs was performed for 60 seconds and/or 10 repetitions.

ELIGIBILITY:
Inclusion Criteria:

* Being >65 years old
* Montreal Cognitive Assessment Scale score > 21
* Diagnosed with Age-Related Hearing Loss
* Having bilateral symmetrical hearing loss (average ±10dB difference)
* Having normal visual functions
* Ability to ambulate independently (may use a self-help device)

Exclusion Criteria:

* Using a hearing aid
* Receiving a physical therapy intervention for Age-Related Hearing Loss
* Having an orthopedic or neurological condition that may affect cognition or postural control
* Using medication that may affect cognition or postural control
* Having vertigo or being hospitalized in the emergency room due to vertigo attacks
* Missing or refusing the follow-up

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Senior Fitness Test | Initially, 1st week
  This test is valid in the elderly population and provides comprehensive, continuous measurement, consisting of 6 sub-heading, including chair stand, arm curl, 2-minute step, chair sit-and-reach, back scratch, and 8-foot-up-and-go tests
Senior Fitness Test | At 5th week
  This test is valid in the elderly population and provides comprehensive, continuous measurement, consisting of 6 sub-heading, including chair stand, arm curl, 2-minute step, chair sit-and-reach, back scratch, and 8-foot-up-and-go tests
Senior Fitness Test | Through study completion at 6th month
  This test is valid in the elderly population and provides comprehensive, continuous measurement, consisting of 6 sub-heading, including chair stand, arm curl, 2-minute step, chair sit-and-reach, back scratch, and 8-foot-up-and-go tests
Montreal Cognitive Assessment | Initially, 1st week
  It evaluates 8 different cognitive functions: visuospatial/executive functions, naming, attention, concentration and calculation, language, abstraction, delayed recall, and orientation. The highest score is 30 in total. A score of 21 and above is considered normal
Montreal Cognitive Assessment | At 5th week
  It evaluates 8 different cognitive functions: visuospatial/executive functions, naming, attention, concentration and calculation, language, abstraction, delayed recall, and orientation. The highest score is 30 in total. A score of 21 and above is considered normal
Montreal Cognitive Assessment | Through study completion at 6th month
  It evaluates 8 different cognitive functions: visuospatial/executive functions, naming, attention, concentration and calculation, language, abstraction, delayed recall, and orientation. The highest score is 30 in total. A score of 21 and above is considered normal
Pure tone audiometry | Initially, 1st week
  Pure tone audiometry at 6 different frequencies (0.5, 1, 2, 4, 6, 8 kHz) frequently mentioned in the literature was performed by an audiologist with a clinical audiometer
World Health Organization Quality of Life - Old Module | Initially, 1st week
  It consists of 24 items in six facets. The facets of this module are "sensory abilities", "autonomy", "past, present and future activities", "social participation", "death and death", "intimacy". A high score indicates a high quality of life.
World Health Organization Quality of Life - Old Module | At 5th week
  It consists of 24 items in six facets. The facets of this module are "sensory abilities", "autonomy", "past, present and future activities", "social participation", "death and death", "intimacy". A high score indicates a high quality of life.
World Health Organization Quality of Life - Old Module | Through study completion at 6th month
  It consists of 24 items in six facets. The facets of this module are "sensory abilities", "autonomy", "past, present and future activities", "social participation", "death and death", "intimacy". A high score indicates a high quality of life.

SECONDARY OUTCOMES:
Berg Balance Scale | Initially, 1st week
  It was designed to assess balance and determine fall risk in older adults (Berg et al, 1989). It is a scale that includes 14 instructions and is scored between 0 and 4 by observing the performance of the person for each instruction. The highest score is 56, 0-20 points indicate balance disorder, 21-40 points indicate that balance is maintained with assistance, and 41-56 points indicate the existence of a good balance
Berg Balance Scale | At 5th week
  It was designed to assess balance and determine fall risk in older adults (Berg et al, 1989). It is a scale that includes 14 instructions and is scored between 0 and 4 by observing the performance of the person for each instruction. The highest score is 56, 0-20 points indicate balance disorder, 21-40 points indicate that balance is maintained with assistance, and 41-56 points indicate the existence of a good balance
Berg Balance Scale | Through study completion at 6th month
  It was designed to assess balance and determine fall risk in older adults (Berg et al, 1989). It is a scale that includes 14 instructions and is scored between 0 and 4 by observing the performance of the person for each instruction. The highest score is 56, 0-20 points indicate balance disorder, 21-40 points indicate that balance is maintained with assistance, and 41-56 points indicate the existence of a good balance
International Fall Efficiency Scale | Initially, 1st week
  : It is a patient-rated scale that determines the level of concerns about falling in activities. of daily living and the confidence to perform activities without fear of falling. It was developed by Tinetti et al. in 1990. The 16 questions in the scale were scored between 1-4. Validity and reliability studies have been established
International Fall Efficiency Scale | At 5th week
  : It is a patient-rated scale that determines the level of concerns about falling in activities. of daily living and the confidence to perform activities without fear of falling. It was developed by Tinetti et al. in 1990. The 16 questions in the scale were scored between 1-4. Validity and reliability studies have been established
International Fall Efficiency Scale | Through study completion at 6th month
  : It is a patient-rated scale that determines the level of concerns about falling in activities. of daily living and the confidence to perform activities without fear of falling. It was developed by Tinetti et al. in 1990. The 16 questions in the scale were scored between 1-4. Validity and reliability studies have been established
Functional Independence Measurement | Initially, 1st week
  FIM was developed in 1987 and it indicates the degree of independence of a person in activities of daily living. The instrument includes 18 items under 6 subheadings: self-care, sphincter control, transfers, locomotion, communication, and social cognition. Each item is scored at 7 levels, with 'level 1' representing full assistance and 'level 7' representing complete independence. The total score is between 18-126.
Functional Independence Measurement | At 5th week
  FIM was developed in 1987 and it indicates the degree of independence of a person in activities of daily living. The instrument includes 18 items under 6 subheadings: self-care, sphincter control, transfers, locomotion, communication, and social cognition. Each item is scored at 7 levels, with 'level 1' representing full assistance and 'level 7' representing complete independence. The total score is between 18-126.
Functional Independence Measurement | Through study completion at 6th month
  FIM was developed in 1987 and it indicates the degree of independence of a person in activities of daily living. The instrument includes 18 items under 6 subheadings: self-care, sphincter control, transfers, locomotion, communication, and social cognition. Each item is scored at 7 levels, with 'level 1' representing full assistance and 'level 7' representing complete independence. The total score is between 18-126.
Dual Task Questionnaire | Initially, 1st week
  : DTQ is used to provide information about the difficulties experienced in dual tasks related to daily living activities. It is a short test consisting of 10 questions. It has been used in patients with stroke and traumatic brain injury. It consists of 5 answers and is scored between 0-4. A score of "4" indicates that difficulties are experienced very often, and "0" indicates that there is no difficulty.
Dual Task Questionnaire | At 5th week
  : DTQ is used to provide information about the difficulties experienced in dual tasks related to daily living activities. It is a short test consisting of 10 questions. It has been used in patients with stroke and traumatic brain injury. It consists of 5 answers and is scored between 0-4. A score of "4" indicates that difficulties are experienced very often, and "0" indicates that there is no difficulty.
Dual Task Questionnaire | Through study completion at 6th month
  : DTQ is used to provide information about the difficulties experienced in dual tasks related to daily living activities. It is a short test consisting of 10 questions. It has been used in patients with stroke and traumatic brain injury. It consists of 5 answers and is scored between 0-4. A score of "4" indicates that difficulties are experienced very often, and "0" indicates that there is no difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: HANDE USTA, PHD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Kinikli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruce H, Lai L, Bherer L, Lussier M, St-Onge N, Li KZH. The effect of simultaneously and sequentially delivered cognitive and aerobic training on mobility among older adults with hearing loss. Gait Posture. 2019 Jan;67:262-268. doi: 10.1016/j.gaitpost.2018.10.020. Epub 2018 Oct 23. PMID 30390596
- [Background] Bruce H, Aponte D, St-Onge N, Phillips N, Gagne JP, Li KZH. The Effects of Age and Hearing Loss on Dual-Task Balance and Listening. J Gerontol B Psychol Sci Soc Sci. 2019 Jan 10;74(2):275-283. doi: 10.1093/geronb/gbx047. PMID 28486677